CLINICAL TRIAL: NCT05247346
Title: Early Detection of Cancer Onset Based on Sensing Field Cancerization at the Organ Level in the Alimentary Tract Using an Integrated Stimulated Raman/Scattering Modality for Endoscopic Real-time in Vivo Measurements
Acronym: SENSITIVE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Collaborators: Technical University of Munich (Other); Universidad Carlos III de Madrid (Unknown); Biomedical Research Foundation of the Academy of Athens (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 202100772
Record Dates: First submitted 2022-01-20; First posted 2022-02-18 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Esophageal Adenocarcinoma; Barrett Esophagus; Colorectal Adenoma; Colorectal Polyp; Colorectal Neoplasms; Colorectal Adenocarcinoma; Carcinogenesis
Keywords: Field cancerization; Raman spectroscopy; Scattering measurements; Surveillance
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Barrett Esophagus; Colorectal Neoplasms; Carcinogenesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- probe-based endoscopic Raman and scattering measurements of GI tissue (Experimental): probe-based integrated Raman spectroscopy and scattering measurements of BE and colorectal tissue during GI endoscopy
  Interventions: Device: SENSITIVE system

INTERVENTIONS:
Device: SENSITIVE system — probe-based integrated Raman spectroscopy and scattering measurements of Barrett's and colorectal tissue during GI endoscopy

SUMMARY:
The investigators hypothesize that detection of field cancerization in the GI tract could be performed during endoscopy by performing Raman and scattering measurements. Together with the Technical University of Munich (TUM) and the Universidad Carlos III de Madrid (UC3M), the investigators have developed an investigational medical device that integrates probe-based Raman and scattering measurements for endoscopic purposes: the SENSITIVE system. During preclinical ex vivo studies, the investigators have established that measurements of the SENSITIVE system were able to discriminate between non-field cancerized tissue and field cancerized tissue. Considering these results, the investigators aim to assess the safety of in vivo Raman/scattering during endoscopy. Secondly, the investigators to assess the feasibility of this approach measurements to determine field cancerization in the alimentary tract during endoscopy through the SENSITIVE system.

DETAILED DESCRIPTION:
Esophageal adenocarcinoma and colorectal carcinoma are common conditions that are responsible for high mortality rates among the worldwide population. Respectively, patients with Barrett's esophagus and Lynch syndrome are known to be at risk of developing these lethal conditions. Therefore, these patients are subject to regular endoscopic surveillance in order to screen for the presence of these malignancies in order to detect the lesions during their premalignant stages. However, the intervals at which these screening examinations have been stratified have an empirical basis with an arbitrary span of time leading to a lot of unnecessary invasive examinations in the majority of these patients. Preferably, a tailored strategy is applied to patients that have an established risk of developing a cancerous lesion. In order to achieve this approach, detection of field cancerization could play a key role. Before histopathological manifestations of disease develop, subtle changes in cells and tissue occur as elements of field cancerization. If these changes can be observed in vivo in real-time, field cancerization can be diagnosed. Subsequently, patients could be more precisely stratified in a in high- and low-risk cohorts and intervals of surveillance examinations could be adapted. Furthermore, if field cancerization would be identified in real-time during endoscopy, it could be used during therapeutic endoscopies for assessment of (residual) tissue. For the detection of field cancerization, advanced biomedical optical techniques that can visualize nanoscale biomarkers are required. Therefore, the investigators developed an integrated Raman/scattering modality that can perform probe-based measurements of the alimentary mucosa during GI endoscopy. Raman spectroscopy provides information regarding the biomolecular composition of the tissue while measuring the scattering properties provides structural information on a nanoscale.

During our preclinical studies, the investigators investigated the feasibility of Raman and scattering measurements for detecting field cancerization on human tissue (BE and colon) samples and tissue samples from murine models (intestinal model: villin-Cre/APCco/wt mice, and BE model: L2-IL1B/WT mice, healthy control models: WT mice). Human biopsies included BE and colorectal samples of non-suspected tissue from organs without an established dysplastic lesion (group A; without expected field cancerization), and non-suspected tissue from organs with an established dysplastic lesion (group B; expected field cancerization). In addition, samples were obtained from dysplastic lesions in BE patients (Group C).

Non-affected human tissue samples from Group B showed remarkably concentered results along the Raman spectrum, which appeared to show more similarity to the Raman results of the dysplastic lesion-samples rather than the other non-affected tissue samples from Group. A. The samples from group A showed a large variability of data along their Raman spectrum. This variability hampered to establish significant differences in the non-affected tissue samples from organs without expected field cancerization to the ones from the organs with expected field cancerization. Interestingly, increases in the three parameters measured by the scattering (disorder strength, depolarization rate, and roughness frequency) were all discriminative for non-affected tissue samples from BEs with established field cancerization (Group B) from the non-affected samples from BEs without expected field cancerization (Group A). In the rectum, solely the disorder parameter yielded significant differences between non-dysplastic colon tissue vs tissue from colons with established field cancerization.

In the murine models that grew EAC and intestinal cancer, the Raman measurements of dysplastic tissue samples showed different peaks of wavenumbers in the Raman spectrum compared to the normal tissue samples of the WT at different organ level (forestomach, SCJ, stomach, intestine). Moreover, Raman results enabled differentiation of non-affected tissue samples from mice with field cancerization (i.e. containing an established tumor) compared to normal/non-affected tissue samples from WT mice (i.e. not to have field cancerization). In addition, the combination of parameters of the scattering and PWS modalities result in a sensitive detection modality that van be used in an auxiliary fashion to the Raman cancer screening.

Thus, the investigators hypothesize that an integrated approach of Raman spectroscopy and scattering measurements enable the detection of field cancerization of esophageal and colorectal tissue.

Therefore, the investigators aim to assess the safety of probe-based scattering and Raman measurements using the SENSITIVE system of alimentary mucosa during GI endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for either a gastroscopy in the context of a Barrett's esophagus or a colonoscopy in the context of colorectal polyps;
* Age of 18 years or older;
* Written informed consent.

Exclusion Criteria:

* Patients with simultaneous neoplasia elsewhere in the GI tract;
* Patients with a medical history of head and neck or lung cancer;
* Patients with a history of endoluminal ablative therapy or radiation therapy;
* Patients younger than 18 years
* Other medical conditions of the esophagus or colon that potentially can disturb measurements of the SRS/scattering spectra such as (eosinophil) esophagitis, inflammatory bowel disease or a medical history of radiation therapy;
* Physical or mental disorders that comprise the ability of the patient to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of intervention-emergent adverse events and serious adverse events | 1 year
  Safety of endoscopic Raman/scattering measurements according to AEs, SAEs, and SUSARs

SECONDARY OUTCOMES:
Raman parameters | 1 year
  Feasibility of the probe-based measurements for the detection of field cancerization
Scattering parameters | 1 year
  Feasibility of the probe-based measurements for the detection of field cancerization

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands